CLINICAL TRIAL: NCT03232229
Title: Supplementation in Tennis: an Observational Study
Brief Title: Supplementation in Tennis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Laurent Chapelle, Researcher, Vrije Universiteit Brussel
Other Study IDs: Suppl Tennis
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Supplements; Tennis; Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tennis players

SUMMARY:
The aim of this observational study is to examine supplementation (e.g. caffeine or creatin) use in both male and female professional tennis players.

ELIGIBILITY:
Inclusion Criteria:

* Professional tennis player

Exclusion Criteria:

* Any metabolic disease or a possible pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants will have to be professional tennis players, both male and female.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Supplementation questionnaire | October 2017 - September 2018
  The participants will be asked about their supplementation use using a questionnaire. Participants will have a list of possible supplements on this questionnaire and they will be asked to indicate which supplement they take on a regular basis (at least once every three months).
  The primary outcome measure will be the frequency (as a percentage) of the supplement intake.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.